CLINICAL TRIAL: NCT05601674
Title: The Effect of Low Flow Anesthesia on Postoperative Emergence Agitation in Rhinoplasty: A Randomized, Controlled Trial
Brief Title: The Effect of Low Flow Anesthesia on Postoperative Emergence Agitation in Rhinoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ülkü Özgül, Professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: Low Flow Anesthesia
Record Dates: First submitted 2022-10-27; First posted 2022-11-01 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Emergence Agitation; Anesthetics; Rhinoplasty
Keywords: Emergence Agitation; Anesthetics
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional group (Placebo Comparator): Anesthesia induction will be performed with 2 mg/kg propofol, 1 µg/kg fentanyl and 0.6 mg/kg rocuronium as standard.After intubation, anesthesia will maintained with %40 O2 and sevoflurane at 2% volume. When the sevoflurane concentration reached 1 MAC, the fresh gas flow rate will be brought to 2 L/min. Inhalation anesthetics will be turned off 10 minutes before the end of the operation. The fresh gas flow will be increased to 6 l/min to be 100% O2. At the end of the surgery, the neuromuscular block will be antagonized with neostigmine-atropine. Sedation and agitation will be assessed immediately after extubation.
  Interventions: Other: : Conventional flow Anesthesia
- Low Flow Group (Active Comparator): anesthesia induction will be performed with 2 mg/kg propofol, 1 µg/kg fentanyl and 0.6 mg/kg rocuronium as standard.After intubation, anesthesia will maintained with %40 O2 and sevoflurane at 2% volume. When the sevoflurane concentration reached 1 MAC, the fresh gas flow rate will be brought to 0.5 L/min. Inhalation anesthetics will be turned off 10 minutes before the end of the operation. The fresh gas flow will be increased to 6 l/min to be 100% O2. At the end of the surgery, the neuromuscular block will be antagonized with neostigmine-atropine. Sedation and agitation will be assessed immediately after extubation.
  Interventions: Other: Low Flow Anesthesia

INTERVENTIONS:
Other: : Conventional flow Anesthesia — During the initial wash-in period 2 L/min Fresh gas flow will be used.
  Arms: Conventional group
Other: Low Flow Anesthesia — Fresh gas flow rate will be 0.5 L/min throughout the procedure.
  Arms: Low Flow Group

SUMMARY:
Emergence agitation, defined as restlessness, disorientation, arousal, and/or inconsolable crying, is a common phenomenon seen in the early phase of recovery from general anesthesia; this may cause respiratory depression, nausea and vomiting, as well as an increase in blood pressure, heart rate and myocardial oxygen consumption. Although its pathogenesis remains unclear, ENT (ear, nose and throat) surgical procedures have been reported to have a higher incidence of agitation in both adults and children. In recent years, low-flow inhalation anesthesia has been widely used in adult anesthesia practice. The aim of this study is to compare the effects of low flow anesthesia and normal flow anesthesia on emergence agitation.

DETAILED DESCRIPTION:
Emergence agitation, defined as restlessness, disorientation, arousal, and/or inconsolable crying, is a common phenomenon seen in the early phase of recovery from general anesthesia; this may cause respiratory depression, nausea and vomiting, as well as an increase in blood pressure, heart rate and myocardial oxygen consumption. Hypoxia can lead to serious complications such as aspiration pneumonia, bleeding or reoperation. Although its pathogenesis remains unclear, ENT (ear, nose and throat) surgical procedures have been reported to have a higher incidence of agitation in both adults and children.

In recent years, low-flow inhalation anesthesia has been widely used in adult anesthesia practice. Low flow anesthesia has many advantages; the consumption of inhalation agents is reduced, the temperature and humidity of the airways are maintained, the cost of anesthesia and pollution caused by atmospheric waste gases are reduced. In addition, because the temperature and humidity of the tracheobronchial tree are preserved, respiratory functions and mucociliary activities are better preserved. In low-flow anesthesia, the concentration of inhaled anesthetics changes very slowly, and their concentration gradually decreases after the administration is terminated. Since the anesthetic concentration will slowly decrease in the low-flow group during termination of anesthesia, the concentration difference between the brain and lungs will be small. In addition, it is known that a longer period between discontinuation of the administration of anesthetic agents and extubation reduces emergence agitation. This seems possible with the low-flow anesthesia technique.

The aim of this study is to compare the effects of low flow anesthesia and normal flow anesthesia on emergence agitation.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years
* ASA class I-II,
* scheduled for elective rhinoplasty surgery under general anesthesia

Exclusion Criteria:

* history of allergy to nonsteroidal anti-inflammatory drugs,
* bleeding diathesis or anticoagulant use,
* psychiatric drug use,
* previous rhinoplasty surgery
* patient refusal

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Richmond Agitation-Sedation Scale (RASS) | From extubation to 30 minutes of arrival in the postoperative care unit
  Sedation and agitation will be assessed immediately after extubation with the Richmond Agitation-Sedation Scale. RASS is divided into 10 levels (score range, -5 to 4, higher scores indicate more agitation)

SECONDARY OUTCOMES:
Ramsey Sedation Scale (RSS) | From extubation to 30 minutes of arrival in the postoperative care unit
  RSS is divided into 6 levels (score range, 1-6, lower scores indicate more agitation).
Boezaart score | immediate postoperative period
  the quality of the operating field in terms of bleeding (Boezaart score),Participating surgeons will rate surgical site visibility from 0 to 5 on the Boezaart rating scale, where 0 is the best and 5 is the worst.
Surgeon satisfaction | immediate postoperative period
  . Surgeon satisfaction with the operative field will be rated at the end of surgery using a 5-choice Likert scale: 1 = very bad, 2 = bad, 3 = fair, 4 = good, and 5 = excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Ulku Ozgul, Professor, Principal Investigator — Inonu University
Locations (1):
- Ulku Ozgul, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yu D, Chai W, Sun X, Yao L. Emergence agitation in adults: risk factors in 2,000 patients. Can J Anaesth. 2010 Sep;57(9):843-8. doi: 10.1007/s12630-010-9338-9. Epub 2010 Jun 5. PMID 20526708